CLINICAL TRIAL: NCT05053984
Title: Ultrasound-Guided Percutaneous Neuromodulation in Spasticity
Acronym: NEUROECO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEUROECO
Record Dates: First submitted 2021-08-26; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuromodulation (Experimental): This study has only 1 arm and the control group is their baseline data
  Interventions: Procedure: Percutaneous Echoguided Neuromodulation

INTERVENTIONS:
Procedure: Percutaneous Echoguided Neuromodulation — Once the nerve is located, a needle is introduced in the vicinity of the nerve and is stimulated using an electrical current with a frequency of 10 Hz, with a pulse width of 250 µs and a tolerable intensity causing a visible muscle contraction for 1.5 minutes.

SUMMARY:
The Multiple sclerosis (MS) is a chronic, inflammatory, autoimmune disease characterised by the appearance of lesions, characterised by heterogeneity in their anatomopathological, clinical and radiological presentation.

Its aetiology is complex and multifactorial, with genetic and environmental interactions with a predominance in women (3:1) and is the second leading cause of disability in young adults (25-30 years). It has a socio-economic impact, affecting interpersonal relationships and causing a significant reduction in quality of life.

MAIN OBJECTIVE To assess the effect on spasticity of the Percutaneous Ultrasound-guided Neuromodulation (PMN) technique in patients diagnosed with MS with upper limb spasticity.

SECONDARY OBJECTIVES

* To assess changes in the strength parameter of the wrist flexor musculature wrist before and after the application of a PMN programme.
* To assess changes in the functionality scales (modified Asworth, established for spasticity
* To assess changes in the range of motion (ROM) of the joints under study.
* Assess changes in the quality of life scale (MSQOL54).
* To assess the adverse effects of the technique.

All patients will receive a Percutaneous Echoguided Neuromodulation (PNM) in the median nerve at the elbow, medial to the brachial artery, running between the humeral and ulnar heads of the pronator teres muscle. Once the nerve is located, a needle shall be inserted in the vicinity of the nerve and is stimulated using an electrical current with a frequency of 10 Hz, with a pulse width of 250 µs and a tolerable intensity causing a visible muscle cont raction for 1.5 minutes.

After assessing the correct application of ethics in the study, it was decided to use the individual's own baseline data as a control group, as simulating the technique is complex.

ELIGIBILITY:
Inclusion Criteria:

* Sign the consent form to participate in the study
* Be a patient diagnosed with Multiple Sclerosis.
* Be over 18 years of age and less than or equal to 55 years of age.
* Have spasticity (Asworth 2) in the upper limb.
* Be able to travel to the place of the session

Exclusion Criteria:

* Failure to comply with the above
* Withdrawal of informed consent
* Having a disease associated with MS that is incompatible with the technique. Use of anticoagulation
* Cognitive impairment
* Belenophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-02 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Spasticity | 8 weeks
  Modified Ashworth Scale which is a measure for the quantification of hypertonia of any articulation. It is a qualitative exam, with values in a range 0 to 4.
Patient's quality of life | 8 weeks
  MSQOL 54: It's a questionnaire that measure mental and physical aspects. The range is from 0 to 100, where 100 is the highest grade of quality of life
Patient Functionality | 8 weeks
  Barthel Index: It's a measure of physical disability which assess functional disability in the activities of the daily life (ADL). The global range can vary between 0 (completely dependent) and 100 points (completely independent)
9 hole peg test | 8 weeks
  9HP: Test to assess limb function upper / hand. The patient is asked to incorporate 9 pins into a board with 9 holes, one in each hole, as fast as they can using their dominant hand. Once the test is done, it is repeated one more time for each hand.
Muscle strength | 8 weeks
  Dynamometer: Dynamometry is an objective way of measuring muscle strength performed by an individual, managing to express it as a quantitative variable, which facilitates its assessment.
Range of Motion | 8 weeks
  Goniometer: Is used to assess changes in the range of motion (ROM) of the joints. The measurements made can be influenced by different factors: the ability to locate appropriate anatomical landmarks, evaluator experience, sex, weight, and age of the subject, as well as the type of joint. the level of reliability in the scan is somewhat greater in the joints of the upper limb than in the lower limb and this rises when more measurements are taken by the same examiner and on the same day.
Satisfaction Scale | Immediately after the treatment
  EVA Scale: It is an instrument for measuring subjective characteristics or attitudes that cannot be measured directly. Range:1-10

CONTACTS AND LOCATIONS:
Locations (1):
- UICEC, San Cristóbal de La Laguna, S/C de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No